CLINICAL TRIAL: NCT07326280
Title: The Impact of Cold Ischemia on Recovery From Ischemia After Robot-assisted Partial Nephrectomy: A Randomized Controlled Clinical Study
Brief Title: The Cold Ischemia Robot-assisted Partial Nephrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SL-B2022-518-03
Record Dates: First submitted 2025-11-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Renal Cell Carcinoma; Renal Function Abnormal
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: Randomly dividing the study cohorts into two groups. One group undergoing cold ischemia robot-assisted partial nephrectomy，while the other group undergoing warm ischemia robot-assisted partial nephrectomy
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold ischemia (Experimental): During the surgical procedure, employing ice to achieve local hypothermia in the kidneys.
  Interventions: Procedure: Cold ischemia robot-assisted partial nephrectomy
- Warm ischemia (Active Comparator): Not applying local hypothermia to the kidneys during the surgical procedure
  Interventions: Procedure: Warm ischemia robot-assisted partial nephrectomy

INTERVENTIONS:
Procedure: Cold ischemia robot-assisted partial nephrectomy — During the surgical procedure, employing ice to achieve local hypothermia in the kidneys.
  Arms: Cold ischemia
Procedure: Warm ischemia robot-assisted partial nephrectomy — Not applying local hypothermia to the kidneys during the surgical procedure
  Arms: Warm ischemia

SUMMARY:
To establish evidence that cold ischemia, achieved through the use of ice slush, can improve the recovery from ischemia on the operated kidney in patients undergoing robot-assisted partial nephrectomy.

DETAILED DESCRIPTION:
Randomly dividing the study cohorts into two groups. One group undergoing cold ischemia partial nephrectomy and the other undergoing warm ischemia partial nephrectomy. Comparing the short-term renal function recovery between the two groups.

ELIGIBILITY:
Inclusion Criteria:

- 18 to 80 years old; 2. Intending to perform robot-assisted partial nephrectomy

Exclusion Criteria:

* Anesthesiologist assessment: Patient unsuitable for general anesthesia;
* Having severe cardiovascular and cerebrovascular diseases;
* horseshoe kidney;
* pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recovery from ischemia | 1-12 months after surgery
  (%GFR saved)/(%parenchymal mass preserved)

SECONDARY OUTCOMES:
surgical duration | Intraoperative
  The duration of the surgery
surgical complications | 1-12 months after surgery
  Intraoperative and postoperative complication incidence rate
The extent of decline in the long-term GFR (month13-24) on the operated kidney compared to the new baseline GFR(months 1-12). | up to 2 years after surgery
  Postoperative short-term GFR(months 1-12) minus long-term GFR(month13-24)

CONTACTS AND LOCATIONS:
Overall Officials: Fangjian Zhou, professor, Principal Investigator — Sun Yat-sen University Cancer Center (SYSUCC)
Locations (1):
- 651 Dongfeng Road East, Yuexiu District, Guangzhou, P.R. China Sun Yat-sen University Cancer Center；, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No